CLINICAL TRIAL: NCT00617747
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Parallel Group Trial to Evaluate Early Efficacy and Tolerability of Zolmitriptan (ZOMIG) Nasal Spray in the Acute Treatment of Adult Subjects With Migraine.
Brief Title: Efficacy and Tolerability of Zolmitriptan Nasal Spray
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 311CUS/0022; D1221L00001
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Migraine
Keywords: Zolmitriptan; ZOMIG; migraine; headache response; headache; headache pain
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — zolmitriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Zolmitriptan
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolmitriptan — 5mg Nasal Spray
  Other Names: Zomig
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability (the ability not to experience ill effects from the study drug) of a zolmitriptan nasal spray, 5.0 mg, compared with placebo (inactive drug) for 2 migraine headaches for up to 12 weeks in adult subjects with migraine headaches

ELIGIBILITY:
Inclusion Criteria:

* Subject has an established diagnosis of migraine headache, with or without aura
* Subject has a medical history indicating the presence of migraine attacks for at least 1 year before the start of the trial or a minimum of 2 and maximum of 6 migraine attacks per month on average for 3 months preceding the study
* Subject has non migraine headaches on fewer than 6 days each month for 3 months preceding the study

Exclusion Criteria:

* Subject has history of basilar, ophthalmoplegic or hemiplegic migraine or serious neurologic condition associated with headache
* Subject has used a MAOI within 2 weeks of randomisation or has been given SSRI therapy or migraine prophylactic agent within 3 months of randomisation. Subject requires treatment with propranolol or cimetidine or has had an intolerable or serious adverse event while using another triptan
* Subject has a history or symptoms suggestive of ischemic heart disease, coronary artery vasospasm or other significant underlying cardiovascular disease or clinically significant abnormalities seen on an ECG or uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2114 (Actual)
Dates: Start 2002-09; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Improvement in migraine headache pain from severe or moderate to mild or none | 15 minutes after the initial dose of trial treatment

SECONDARY OUTCOMES:
Headache response rate | 30 minutes and 1, 2 and 4 hours after dosing